CLINICAL TRIAL: NCT04234165
Title: Safety and Efficacy of Bipolar vs Monopolar Transurethral Resection of Bladder Tumor-A
Brief Title: Safety and Efficacy of Bipolar vs Monopolar Transurethral Resection of Bladder Tumor-A Randomized Controlled Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tribhuvan University, Nepal (Other)
Responsible Party: Principal Investigator, Manish Pradhan, Urology Lectuerer, Tribhuvan University, Nepal
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 344-(6-11-E)073-074
Record Dates: First submitted 2020-01-09; First posted 2020-01-21 (Actual); Last update posted 2020-01-21 (Actual); Status verified 2020-01

CONDITIONS: Obturator Jerk in TURBT

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Monopolar arm (Active Comparator): monopolar cautery was used for TURBT
  Interventions: Device: TURBT
- Bipolar Arm (Experimental): bipolar cautery was used for TURBT
  Interventions: Device: TURBT

INTERVENTIONS:
Device: TURBT — different power sources ( bipolar vs monopolar)

SUMMARY:
Study design:

This was a single center, parallel arm, randomized, controlled trial done at Tribhuvan University Teaching Hospital,Institute Of Medicine from May 2017 to April 2018. The allocation ratio was 1:1.

Inclusion criteria: All patients undergoing Transurethral Resection of Bladder Tumor for suspected bladder tumors.

Exclusion criteria were: Consent withdrawal, bladder tumour other than in the lateral wall, unfit for spinal anesthesia and need of general anesthesia or obturator nerve block.

Methodology:

All patients suspected to have bladder cancer were subjected to imaging or cystoscopy and with confirmation of the diagnosis; they were randomized into two arms of TURBT. Spinal anesthesia was used in all cases. To overcome the potential confounding effect on our primary end point, obturator jerk, nerve block was not used.

Cystoscopy was done first and the findings were noted before proceeding to TURBT.

Tumors were resected in block from periphery to center with the stalk resected last. An additional sample of deep muscle was obtained from the tumor base and sent for histopathological examination in different containers.

All study variables were recorded in Per forma during the operation and in post operative period. Hemoglobin and sodium level was determined in immediate post operative period.

Postoperative irrigation was done with normal saline in both the resection groups and continued till the urine was clear. The catheter was removed after 48 hours in uncomplicated cases and patients were discharged. Patients were followed up in OPD at 2 weeks with the

DETAILED DESCRIPTION:
All patients suspected to have bladder cancer were subjected to imaging or cystoscopy and with confirmation of the diagnosis; they were randomized into two arms of TURBT. Spinal anesthesia was used in all cases.

To overcome the potential confounding effect on our primary end point, obturator jerk, nerve block was not used.

Cystoscopy was done first and the findings were noted before proceeding to TURBT.

Monopolar resection was done using 1.5% Glycine solution at 110 watt cutting, and 70 watt coagulation power (Covidien Valley-lab Force Fx TM) with Karl Storz 26f resectoscope and loop (8mm width and 5mm depth) with 300 telescope. Bipolar resection was done with 0.9% Normal Saline with digital impedence dependent cutting (power range 150-250 watt) and 80 watt coagulation power (Bowa Arc 400) with Karl Storz 26f resectoscope and loop (6mm width and 5mm depth) with 300 telescope.

Tumors were resected in block from periphery to center with the stalk resected last. An additional sample of deep muscle was obtained from the tumor base and sent for histopathological examination in different containers. All study variables were recorded in Per forma during the operation and in post operative period. Hemoglobin and sodium level was determined in immediate post operative period.

Postoperative irrigation was done with normal saline in both the resection groups and continued till the urine was clear. The catheter was removed after 48 hours in uncomplicated cases and patients were discharged. Patients were followed up in Out Patient Department at 2 weeks with the histopathological report for or when necessary.

Study outcome:

The incidence of obturator jerk, bladder perforation, resection time, decrease in hemoglobin and serum sodium, clot retention, need for blood transfusion, need for recoagulation and TUR syndrome were recorded for the cases in both arms. All resected specimen were evaluated by pathologist for quality by determining the presence of deep muscle in the sample and comparing the degree of cautery artifact. Severe artifact was defined as more than 50% cautery artifact in most chips.

Statistical Analysis:

Sample size (n) was calculated using 80% power and a 95% significance level for obturator jerk, assuming a 30% incidence for the monopolar system and a 5% incidence for the bipolar system. These values were arrived at after a comprehensive literature review. The sample size was determined with the formula n= K {P1(1-P1) x P2(1-P2)}/ )P1-P2)2, Where:

N= sample size P1= prevalence of obturator jerk in Monopolar TURBT P2= prevalence of obturator jerk in Bipolar TURBT K= constant (7.9 for 80% power of study and 0.05 level of significance)

A sample size of 33 in each arm was calculated using above formula. Estimating a drop out of 10%, we decided to include at least 37 patients in each arm. A computer generated random number was used to allocate eligible patients in to monopolar or bipolar resection arm. Data analysis was done using Statistical Package for Social Sciences (SPSS) version 21. Significance was determined using the independent sample t-test for quantitative variables and the chi-square test for qualitative data. P value of <0.05 was considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* All patients undergoing TURBT for suspected bladder tumors.

Exclusion Criteria:

* Consent withdrawal, bladder tumour other than in the lateral wall, unfit for spinal anesthesia and need of general anesthesia or obturator nerve block.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2017-05-01 (Actual); Primary Completion 2018-04-01 (Actual); Study Completion 2018-11-01 (Actual)

PRIMARY OUTCOMES:
obturator jerk occurrence | during TURBT
  occurrence of obturator jerk (yes/no) will be recorded

SECONDARY OUTCOMES:
bladder perforation(yes/no) | during TURBT
  this parameter will be recorded during operation
time of resection (minutes | during TURBT
  this parameters will be recorded during operation
TUR syndrome (yes/no) | during and after operation
  this parameters will be recorded during and after operation
decrease in hemoglobin (mg/dl) | immediate post operative period
  this parameters will be recorded immediately after operation
serum sodium(meq/l) | immediate post operative period
  this parameters will be recorded immediately after operation
need for blood transfusion (yes/no) | immediate post operative period
  this parameters will be recorded immediately after operation
clot retention (yes/no) | immediate post operative period
  this parameters will be recorded immediately after operation
presence of deep muscle (yes/no) | two weeks after operation ( as per usual availability of histopathology report in the hospital)
  histo-pathology report will be evaluated for these outcome
severy cautery artifact(yes/no) | two weeks after operation ( as per usual availability of histopathology report in the hospital)
  histo-pathology report will be evaluated for these outcome

CONTACTS AND LOCATIONS:
Locations (1):
- TUTH, Kathmandu, Three, Nepal

IPD SHARING:
Plan to Share IPD: Yes
online availability
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code